CLINICAL TRIAL: NCT04125134
Title: Predicting the Success of Dry Eye Disease Interventions Using Clinical Tests
Acronym: PreDICT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties (low accrual)
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13363
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye
Keywords: Dry Eye; artifical tear
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hypertonic Saline Responders (Experimental): Subjects who qualify as hypertonic saline responders will be instructed to instill 1-2 drops of preservative-free Refresh Optive Advanced Lubricant Eye Drops, which are available over the counter, into each eye twice a day for 28 days.
  Interventions: Drug: Preservative-free Refresh Optive Advanced Lubricant Eye Drops
- Hypertonic Saline Non-responders (Experimental): Subjects who qualify as hypertonic saline non-responders will be dispensed the same instructions and treatment as the Hypertonic Saline Responders. They will be instructed to instill 1-2 drops of preservative-free Refresh Optive Advanced Lubricant Eye Drops, which are available over the counter, into each eye twice a day for 28 days.
  Interventions: Drug: Preservative-free Refresh Optive Advanced Lubricant Eye Drops

INTERVENTIONS:
Drug: Preservative-free Refresh Optive Advanced Lubricant Eye Drops — over the counter artificial tear

SUMMARY:
This is a single site, prospective, cross-sectional, controlled clinical study on a total of 66 subjects. The subjects are divided into two groups: Hypertonic Saline Non-Responders (33 subjects) and Hypertonic Saline Responders (33 subjects). After completion of questionnaires, the subjects will undergo Dry Eye Disease testing and functional nerve testing. Subjects who qualify will be dispensed 4 weeks of preservative free artificial tears and instructed to instill one drop into each eye twice daily. Subjects will return for a follow up visit 4 weeks later (± 4 days), during which subjects will complete the questionnaires again and the Dry Eye Disease tests and functional nerve tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Hypertonic saline non-responders):

* At least 18 years of age
* Ability to consent
* Diagnosis of Dry Eye Disease (DED) based on:

  * Symptoms of DED, shown with SANDE score of 50mm or greater
  * Two or more of the following objective signs in the same eye: 1. Schirmer test of 10 mm or less over 5 minutes; 2. Fluorescein tear break-up time (FTBUT) of 7 seconds or less; 3. Meibomian gland expression (MGE) grade of 2 or greater for at least 3 out of 5 glands
* HS response result of one of the following:

  * Reduction of discomfort/pain rating
  * No change of discomfort/pain rating
  * Increase in discomfort/pain rating score of 1 step or less

Group 2 (Hypertonic saline non-responders):

* At least 18 years of age
* Ability to consent
* Diagnosis of DED based on:

  * Symptoms of DED, shown with SANDE score 50mm or greater
  * Two or more of the following objective signs in the same eye: 1. Schirmer test of 10 mm or less over 5 minutes; 2. Fluorescein tear break-up time (FTBUT) of 7 seconds or less; 3. Meibomian gland expression (MGE) grade of 2 or greater for at least 3 out of 5 glands
* HS response result of an increase in discomfort/pain rating of greater than 1 step

Exclusion Criteria:

* Presence of centralized pain as indicated by a proparacaine challenge test (PCT) of less than 50% ocular surface discomfort reduction
* Unable to speak English
* History of ocular surgery, corneal infection, or corneal injury within the last 3 months
* Active ocular allergies or other condition that could impact the study results
* Allergic to benzalkonium chloride "BAK" (an eye-drop preservative)
* Changes in topical or systemic medications in the last 3 months or anticipated changes in medication during the course of treatment
* Use of other topical treatments
* Concurrent enrollment in other studies that in the opinion of the investigator will interfere with the results of this study
* Use of contact lenses within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in SANDE severity score response from visit 1 to visit 2 | 4 weeks
  The SANDE questionnaire is a paper and pencil questionnaire consisting of two questions (1. severity of dry eye disease symptoms and 2. frequency of dry eye disease symptoms), which are answered on a continuous visual analogue scale. The severity response from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.

SECONDARY OUTCOMES:
Change in tear break up time from visit 1 to visit 2 | 4 weeks
  The tear break up time is a measure of the stability of the tear film. The measurement from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.
Change in Schirmer test from visit 1 to visit 2 | 4 weeks
  The Schirmer test is a measure of tear production. The measurement from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.
Change in meibomian gland expression from visit 1 to visit 2 | 4 weeks
  Meibomian gland expression allows for a measure of the health of the meibomian glands. The measurement from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.
Change in proparacaine challenge test from visit 1 to visit 2 | 4 weeks
  The proparacaine challenge test allows for a measure of the amount of peripheral neuropathic pain compared to centralized neuropathic pain. The measurement from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.
Change in hypertonic saline response test from visit 1 to visit 2 | 4 weeks
  The hypertonic saline response is expected to be able to assess the severity of dry eye disease. The measurement from visit 2 will be subtracted from that given in visit 1 to provide a subject change. The results of those in the hypertonic saline response group will be compared to those within the hypertonic non-response group.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cox, OD, Principal Investigator — Tufts Medical Center New England Eye Center
Locations (1):
- Tufts Medical Center-New England Eye Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Belmonte C, Aracil A, Acosta MC, Luna C, Gallar J. Nerves and sensations from the eye surface. Ocul Surf. 2004 Oct;2(4):248-53. doi: 10.1016/s1542-0124(12)70112-x. PMID 17216099
- [Background] Shaheen BS, Bakir M, Jain S. Corneal nerves in health and disease. Surv Ophthalmol. 2014 May-Jun;59(3):263-85. doi: 10.1016/j.survophthal.2013.09.002. Epub 2014 Jan 23. PMID 24461367
- [Background] Oliveira-Soto L, Efron N. Morphology of corneal nerves using confocal microscopy. Cornea. 2001 May;20(4):374-84. doi: 10.1097/00003226-200105000-00008. PMID 11333324
- [Background] Tepelus TC, Chiu GB, Huang J, Huang P, Sadda SR, Irvine J, Lee OL. Correlation between corneal innervation and inflammation evaluated with confocal microscopy and symptomatology in patients with dry eye syndromes: a preliminary study. Graefes Arch Clin Exp Ophthalmol. 2017 Sep;255(9):1771-1778. doi: 10.1007/s00417-017-3680-3. Epub 2017 May 20. PMID 28528377
- [Background] Labbe A, Liang Q, Wang Z, Zhang Y, Xu L, Baudouin C, Sun X. Corneal nerve structure and function in patients with non-sjogren dry eye: clinical correlations. Invest Ophthalmol Vis Sci. 2013 Aug 1;54(8):5144-50. doi: 10.1167/iovs.13-12370. PMID 23833066
- [Background] Villani E, Magnani F, Viola F, Santaniello A, Scorza R, Nucci P, Ratiglia R. In vivo confocal evaluation of the ocular surface morpho-functional unit in dry eye. Optom Vis Sci. 2013 Jun;90(6):576-86. doi: 10.1097/OPX.0b013e318294c184. PMID 23670123
- [Background] Labbe A, Alalwani H, Van Went C, Brasnu E, Georgescu D, Baudouin C. The relationship between subbasal nerve morphology and corneal sensation in ocular surface disease. Invest Ophthalmol Vis Sci. 2012 Jul 24;53(8):4926-31. doi: 10.1167/iovs.11-8708. PMID 22695962
- [Background] Benitez-Del-Castillo JM, Acosta MC, Wassfi MA, Diaz-Valle D, Gegundez JA, Fernandez C, Garcia-Sanchez J. Relation between corneal innervation with confocal microscopy and corneal sensitivity with noncontact esthesiometry in patients with dry eye. Invest Ophthalmol Vis Sci. 2007 Jan;48(1):173-81. doi: 10.1167/iovs.06-0127. PMID 17197530
- [Background] Kheirkhah A, Dohlman TH, Amparo F, Arnoldner MA, Jamali A, Hamrah P, Dana R. Effects of corneal nerve density on the response to treatment in dry eye disease. Ophthalmology. 2015 Apr;122(4):662-8. doi: 10.1016/j.ophtha.2014.11.006. Epub 2014 Dec 24. PMID 25542519
- [Background] Mandahl A. Hypertonic saline test for ophthalmic nerve impairment. Acta Ophthalmol (Copenh). 1993 Aug;71(4):556-9. doi: 10.1111/j.1755-3768.1993.tb04636.x. PMID 8249592
- [Background] Rahman M, Okamoto K, Thompson R, Bereiter DA. Trigeminal pathways for hypertonic saline- and light-evoked corneal reflexes. Neuroscience. 2014 Sep 26;277:716-23. doi: 10.1016/j.neuroscience.2014.07.052. Epub 2014 Jul 31. PMID 25086311
- [Background] Yorek MS, Davidson EP, Poolman P, Coppey LJ, Obrosov A, Holmes A, Kardon RH, Yorek MA. Corneal Sensitivity to Hyperosmolar Eye Drops: A Novel Behavioral Assay to Assess Diabetic Peripheral Neuropathy. Invest Ophthalmol Vis Sci. 2016 May 1;57(6):2412-9. doi: 10.1167/iovs.16-19435. PMID 27145474
- [Background] Parra A, Gonzalez-Gonzalez O, Gallar J, Belmonte C. Tear fluid hyperosmolality increases nerve impulse activity of cold thermoreceptor endings of the cornea. Pain. 2014 Aug;155(8):1481-1491. doi: 10.1016/j.pain.2014.04.025. Epub 2014 Apr 28. PMID 24785271
- [Background] Nichols KK, Bacharach J, Holland E, Kislan T, Shettle L, Lunacsek O, Lennert B, Burk C, Patel V. Impact of Dry Eye Disease on Work Productivity, and Patients' Satisfaction With Over-the-Counter Dry Eye Treatments. Invest Ophthalmol Vis Sci. 2016 Jun 1;57(7):2975-82. doi: 10.1167/iovs.16-19419. PMID 27273596
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Qazi Y, Hurwitz S, Khan S, Jurkunas UV, Dana R, Hamrah P. Validity and Reliability of a Novel Ocular Pain Assessment Survey (OPAS) in Quantifying and Monitoring Corneal and Ocular Surface Pain. Ophthalmology. 2016 Jul;123(7):1458-68. doi: 10.1016/j.ophtha.2016.03.006. Epub 2016 Apr 16. PMID 27089999
- [Background] Schaumberg DA, Gulati A, Mathers WD, Clinch T, Lemp MA, Nelson JD, Foulks GN, Dana R. Development and validation of a short global dry eye symptom index. Ocul Surf. 2007 Jan;5(1):50-7. doi: 10.1016/s1542-0124(12)70053-8. PMID 17252166